CLINICAL TRIAL: NCT02761473
Title: Cutaneous Mastocytosis in Children: Analysis of Somatic and Germline Mutations
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1608M92621
Record Dates: First submitted 2016-03-15; First posted 2016-05-04 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Urticaria Pigmentosa; Cutaneous Mastocytosis
MeSH Terms: conditions — Urticaria Pigmentosa; Mastocytosis, Cutaneous | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Buccal swabs, skin biopsy and blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Urticaria Pigmentosa: This group will undergo skin biopsy, blood and buccal swab analyses
  Interventions: Other: skin biopsy; Other: blood draw
- Family members of affected patients: This group will undergo blood and buccal swab analyses

INTERVENTIONS:
Other: skin biopsy — A skin biopsy will be obtained from a typical UP lesion in affected patients
  Groups: Patients with Urticaria Pigmentosa
Other: blood draw — Blood will be obtained from subjects, parents and unaffected siblings
  Groups: Patients with Urticaria Pigmentosa

SUMMARY:
Pediatric mastocytosis is an orphan disease, which encompasses several clinically distinct entities including solitary mastocytoma, urticaria pigmentosa, diffuse cutaneous mastocytosis and the newly recognized mast cell activation syndrome. The most common form of pediatric mastocytosis is cutaneous maculopapular mastocytosis (CMPM), also known as urticaria pigmentosa (UP). There are significant knowledge gaps regarding the genetic basis of pediatric mastocytosis and the functional activity of mast cells in this condition. The Pediatric Dermatology and Pediatric Oncology services at the University of Minnesota Masonic Children's Hospital are seeing significant growth in clinical volumes of pediatric mastocytosis, including rare, familial cases. The aims of this study are to prospectively explore germline risk for UP and to perform a mutational analysis to identify somatic mutations, beyond those currently identified, in pediatric patients with UP.

DETAILED DESCRIPTION:
Urticaria pigmentosa (UP) is a relatively common disorder in pediatric patients, and little is known regarding the somatic and germline genetic variants associated with the disease. The University of Minnesota Masonic Children's Hospital is a regional referral center for pediatric patients with mast cell disorders. Collaborators on this study include several University departments including: Pediatric Dermatology, Pediatric Oncology, the Biomedical Genomics program, Lab Medicine and Pathology department. We hypothesize that because of differences observed in the clinical behavior of pediatric- and adult-onset mast cell disease, specifically UP, we will identify novel somatic gene variants in addition to c-KIT . We further hypothesize that we will observe novel germline genetic variants in pediatric UP distinct from what has previously been described in adults.

Specific Aims include the following:

Specific Aim 1: RNA Sequencing for Gene Expression and Mutation Analysis. Utilizing RNA sequencing (RNA-Seq), we will perform paired lesional and peripheral blood sequencing in UP cases to identify variation in gene expression and define novel somatic mutations associated with pediatric UP.

Specific Aim 2: Exploration of Germline Risk. Utilizing single nucleotide polymorphism (SNP) array, we will perform linkage analysis in UP cases and their unaffected family members to identify germline genetic variants associated with UP.

1. Discordant sibling analysis: Children with UP and their unaffected siblings will be compared to identify germline variants.
2. Identical twin and parent analysis: Identical infant twins with a severe UP phenotype will be compared with their unaffected parents.

ELIGIBILITY:
Inclusion Criteria:

Affected subject:

Subjects will be eligible to participate in the study if all of the following conditions exist:

1. Clinical diagnosis of urticaria pigmentosa/cutaneous mastocytosis with representative skin lesions
2. Age <23 years
3. Capable of giving consent if 18 or older

Inclusion Criteria for Parent:

1. Over 16 years of age
2. Biologic parent to affected subject
3. Capable of providing consent

Inclusion Criteria for Sibling:

1. Biologic sibling to affected subject 2. Capable of giving consent if 18 or older

-

Exclusion Criteria:

1. Absence of skin findings representative of classic urticaria pigmentosa
2. Patients with primarily systemic mastocytosis
3. Unable or unwilling to participate in study procedures

Exclusion Criteria for Parent/Sibling:

1. Unable or unwilling to participate in study procedures

Ages: 3 Months to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients with urticaria pigmentosa and first degree relatives
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
RNA sequencing | 1.5 years
  Fresh tissue from lesional skin will be obtained for gene expression and mutational analysis

SECONDARY OUTCOMES:
SNP microarray analysis | 1.5 years
  SNP microarray analysis will be performed on DNA obtained from buccal swabs or whole blood samples. Samples from patients and unaffected family members will be compared.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hartmann K, Escribano L, Grattan C, Brockow K, Carter MC, Alvarez-Twose I, Matito A, Broesby-Olsen S, Siebenhaar F, Lange M, Niedoszytko M, Castells M, Oude Elberink JNG, Bonadonna P, Zanotti R, Hornick JL, Torrelo A, Grabbe J, Rabenhorst A, Nedoszytko B, Butterfield JH, Gotlib J, Reiter A, Radia D, Hermine O, Sotlar K, George TI, Kristensen TK, Kluin-Nelemans HC, Yavuz S, Hagglund H, Sperr WR, Schwartz LB, Triggiani M, Maurer M, Nilsson G, Horny HP, Arock M, Orfao A, Metcalfe DD, Akin C, Valent P. Cutaneous manifestations in patients with mastocytosis: Consensus report of the European Competence Network on Mastocytosis; the American Academy of Allergy, Asthma & Immunology; and the European Academy of Allergology and Clinical Immunology. J Allergy Clin Immunol. 2016 Jan;137(1):35-45. doi: 10.1016/j.jaci.2015.08.034. Epub 2015 Oct 21. PMID 26476479
- [Result] Longley BJ Jr, Metcalfe DD, Tharp M, Wang X, Tyrrell L, Lu SZ, Heitjan D, Ma Y. Activating and dominant inactivating c-KIT catalytic domain mutations in distinct clinical forms of human mastocytosis. Proc Natl Acad Sci U S A. 1999 Feb 16;96(4):1609-14. doi: 10.1073/pnas.96.4.1609. PMID 9990072
- [Result] Fried AJ, Akin C. Primary mast cell disorders in children. Curr Allergy Asthma Rep. 2013 Dec;13(6):693-701. doi: 10.1007/s11882-013-0392-6. PMID 24150753
- [Result] Fett NM, Teng J, Longley BJ. Familial urticaria pigmentosa: report of a family and review of the role of KIT mutations. Am J Dermatopathol. 2013 Feb;35(1):113-6. doi: 10.1097/DAD.0b013e31826330bf. PMID 22892471